CLINICAL TRIAL: NCT07142863
Title: Single-arm Prospective Clinical Study of PD-L1 Antibody Envafolimab Combined With Neoadjuvant Chemotherapy in Patients With Stage IIb Resectable Osteosarcoma
Brief Title: Envafolimab Combined With Neoadjuvant Chemotherapy Treat Stage IIb Resectable Osteosarcoma Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Mengxiong Sun, Principal Investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024SQ009
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Osteosarcoma; Neoadjuvant Therapy; Neoadjuvant Chemotherapy; PD-L1 Antibody; Envafolimab
MeSH Terms: conditions — Osteosarcoma | interventions — envafolimab; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab combined with neoadjuvant chemotherapy (Experimental)
  Interventions: Drug: Envafolimab and neoadjuvant chemotherapy

INTERVENTIONS:
Drug: Envafolimab and neoadjuvant chemotherapy — * PD-L1 inhibitor envafolimab Paediatric (<18 years): 2.5 mg/kg (maximum 200 mg) by subcutaneous injection on Day 1 of every week (q1w).
  Adult (≥18 years): 200 mg flat dose by subcutaneous injection on Day 1 of every week (q1w).
  * Neoadjuvant chemotherapy--MAP regimen (paediatric patients) Doxorubicin 75 mg/m² intravenously on Days 1-2, administered in weeks 1 and 6 of each 6-week cycle.
  Cisplatin 120 mg/m² intravenously on Days 1-3, administered in weeks 1 and 6 of each 6-week cycle.
  Methotrexate 8-12 g/m² intravenously on Day 1 of weeks 3 and 4 of each 6-week cycle.
  * Neoadjuvant chemotherapy--DIA regimen (adult patients) Doxorubicin 75 mg/m² intravenously on Days 1-2, administered in weeks 1 and 6 of each 6-week cycle.
  Cisplatin 120 mg/m² intravenously on Days 1-3, administered in weeks 1 and 6 of each 6-week cycle.
  Ifosfamide 12-15 g/m² total dose intravenously on Days 1-5 of week 3 of each 6-week cycle.

SUMMARY:
Given that osteosarcoma typically presents at an early age and predominantly affects pediatric and adolescent populations, early control of disease progression and the opportunity for complete tumor resection are particularly crucial. Postoperatively, patients can regain functional mobility through prosthetic implantation and artificial joint reconstruction, thereby preventing premature loss of mobility in young patients. This study aims to explore the efficacy and safety of neoadjuvant treatment with the PD-L1 antibody envafolimab in combination with standard chemotherapy in patients with resectable stage IIb osteosarcoma, and to assess whether this combined regimen can increase the proportion of patients achieving complete tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participate in the study and have good compliance, signing a written informed consent form before enrollment.
* Age between 12 and 70 years, with no gender restrictions.
* Patients diagnosed with non-metastatic, resectable osteosarcoma by pathology and clinical physician assessment.
* Have measurable disease (according to RECIST 1.1 criteria, non-nodal lesions with a CT scan longest diameter ≥10 mm, and nodal lesions with a CT scan shortest diameter ≥15 mm).
* No prior systemic anti-tumor treatment.
* ECOG PS score: 0 to 1.
* Adequate organ function:

  1. Hematological parameters: Absolute Neutrophil Count (ANC) ≥1.5×10^9/L, Platelet (PLT) ≥70×10^9/L, Hemoglobin (HGB) ≥90 g/L.
  2. Hepatic function: Total Bilirubin (TBIL) ≤1.5×Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate Transferase (AST) ≤3×ULN; Serum Albumin ≥28 g/L; Alkaline Phosphatase (ALP) ≤5×ULN; patients on routine hepatic protection treatment meeting the above criteria and stable for at least one week after investigator assessment may be included.
  3. Renal function: Creatinine (Cr) ≤1.5×ULN, or Creatinine clearance rate ≥50 mL/min (using the standard Cockcroft-Gault formula).
  4. Coagulation function: International Normalized Ratio (INR) ≤1.5, Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN; if the subject is undergoing anticoagulant therapy, PT and INR within the intended range of the anticoagulant therapy is acceptable.

Exclusion Criteria:

* Participants with a history of or concurrent diagnosis of other malignant tumors (except for cured cutaneous basal cell carcinoma and in situ cervical carcinoma).
* Patients with recurrent postoperative or previously treated osteosarcoma with local or systemic anti-tumor therapy, or with metastasis.
* Participants who have received the following treatments within 4 weeks prior to study initiation: radiation therapy for tumors, surgical procedures, chemotherapy, immunotherapy, or other investigational drugs.
* Known allergies to any component of the study medication in participants. Participants with uncontrolled clinical symptoms or diseases of the heart, such as: (1) NYHA Class II or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within the past year, (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
* Participants with active infections or fever of unknown origin >38.5°C (measured in Celsius) during the screening period or before the first dose of study medication (fever due to tumors may be included at the discretion of the investigator).
* Use of immunosuppressive drugs within 14 days prior to treatment initiation, excluding intranasal and inhaled corticosteroids or physiological doses of systemic corticosteroids (i.e., daily dose of prednisone ≤10 mg or equivalent physiological doses of other corticosteroids).
* History of active autoimmune diseases or a history of autoimmune disorders (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary glanditis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; participants with vitiligo or asthma that may be in complete remission in childhood and currently do not require medical intervention, or history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation).
* Participants who have received live vaccines within 4 weeks prior to study medication or are likely to receive live vaccines during the study period.
* Participants with a history of substance abuse, alcoholism, or drug addiction.
* Participants deemed to be excluded from this study by the investigator, such as those with other factors that could potentially lead to premature termination of the study, such as other serious diseases (including psychiatric diseases) requiring concomitant treatment, severe laboratory abnormalities, or family or social factors that could affect participant safety, or collection of data and samples.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Tumor necrosis rate | From enrollment to the end of surgery, about 12th weeks.
  According to the Huvos grading system, patient bone tumor specimens were evaluated and analyzed block by block in comparison with preoperative imaging data after sampling, and the data were then summarized. Tumors with necrosis rates of grade I-II were considered to have poor chemotherapeutic response (indicating poor long-term prognosis, and postoperative adjuvant chemotherapy should increase the dose intensity or modify the chemotherapy regimen), while those with necrosis rates of grade III-IV were considered to have a good chemotherapeutic response (it is recommended that postoperative adjuvant chemotherapy use the same chemotherapy regimen as preoperatively). The number of patients in each grade of tumor necrosis rate was counted, and the percentage of patients with tumor cell necrosis rate >90% (i.e., tumor necrosis rate grade III-IV) among all patients will be used as the primary outcome measure.

SECONDARY OUTCOMES:
EFS (event-free survival) | About 1 year.
  The time from the start of treatment to the first occurrence of any of the following events: disease progression precluding the possibility of surgical treatment, local or distant recurrence, or death from any cause.
PFS (Progression-free survival) | About 1 year.
  The time from the start of treatment to disease progression or death of the patient due to any cause.
Immune Microenvironment | About 10th weeks after the start of neoadjuvant therapy (at definitive surgery).
  The immune microenvironment was assessed by single-cell RNA sequencing (scRNA-seq) of surgically resected specimens. The specific measurement is the relative abundance (percentage) of major immune-cell subsets-CD8+ T cells, CD4+ T cells, regulatory T cells (Treg), natural killer (NK) cells, M1 macrophages, and M2 macrophages-within the total viable tumor-infiltrating leukocytes (CD45+ cells) at the time of surgery. Changes in these cell-type proportions between pre-treatment biopsy and post-treatment surgical samples were computed to evaluate the impact of neoadjuvant immune therapy on the tumor microenvironment.
Adverse Events (AEs) | Adverse events (AEs) were recorded after enrollment and within 30 days of the last dose. Serious adverse events or adverse events related to the PD-L1 antibody envafolimab were extended to 90 days after the end of treatment.
  Adverse Events (AEs) according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First People's Hospital, 100 Haining Road, Hongkou District, Shanghai, China

IPD SHARING:
Plan to Share IPD: No